CLINICAL TRIAL: NCT05119985
Title: Ultrasound Guided Peripheral Venous Cannulation in Patient Undergoing Elective Surgery Under General Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Michal Kalina, MUDr., Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: USG kanylace pžk
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Vein Cannulation Guided by Ultrasound
Keywords: ultrasound; vein; cannulation
MeSH Terms: interventions — Catheterization; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Participants are divided by block randomization into two arms. Arm A peripheral vein cannulation with ultrasound guidance and Arm B conventional cannulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound guided cannulation (Active Comparator): Ultrasound guided insertion of peripheral vein cannula.
  Interventions: Procedure: Peripheral vein cannulation
- Cannulation without ultrasound (Active Comparator): Catheter insertion by conventional approach, without ultrasound guidance
  Interventions: Procedure: Cannulation without ultrasound

INTERVENTIONS:
Procedure: Peripheral vein cannulation — The target vein is directly identified by ultrasound, the procedure of peripheral venous catheter insertion is performed conventionally, without ultrasound guidance
  Arms: Ultrasound guided cannulation
Procedure: Cannulation without ultrasound — Cannulation is done the conventional way without any ultrasound use.
  Arms: Cannulation without ultrasound

SUMMARY:
This study evaluates two different techniques for peripheral venous cannulation in operating theatre. Ultrasound guided insertion of peripheral cannula in comparison with conventional approach without any ultrasound guidance.

DETAILED DESCRIPTION:
Peripheral venous catheter placement is one of the key tasks of an anesthesiologist, which needs to be completed before surgery in general anesthesia. The reported success rate of peripheral venous cannulation, when performed in a conventional manner, without any special technical tools which facilitate finding the peripheral vein, is only 51% during the first trial. However, up to 7% of patients require more than three cannulation trials. Ultrasound guidance of peripheral venous catheter insertion may increase success rate and shorten time to securing peripheral cannula. However, this approach has not been verified in the setting of operating theatre so far. This project aims to set the role of ultrasound guided venous cannulation in operating theatre.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years

Exclusion Criteria:

* Age <18 years
* Patient disagreement with the insertion of peripheral venous catheter
* Disagreement of the patient with inclusion in a clinical trial
* Contraindication of ultrasound examination of the venous system
* Contraindication of the introduction of peripheral venous cannula on both upper limbs
* Necessity of securing other vein access than peripheral
* Contraindications of cannulation of peripheral vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Successful Securing of Peripheral Vein on First Attempt | 60 minutes
  Comparing success rate of securing peripheral vein for first attempt in both methods.

SECONDARY OUTCOMES:
Number of Needed Attempts to Successful Securing of Peripheral | 60 minutes
  Compare number of attempts that was necessary to secure peripheral vein.
Number of Complication After and During Securing Peripheral Vein | 24 hours
  Compare complication rate after securing peripheral vein with both methods.
Time Needed to Secure Peripheral Vein | 60 minutes
  Compare time that was need to secure peripheral vein in both methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Masarykova Nemocnice v Ústí nad Labem, Krajská Zdravotní a.s., Ústí nad Labem, Ústí Nad Labem Region, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736